CLINICAL TRIAL: NCT03603080
Title: A Prospective Randomized Study Evaluating the Efficacy of Pharmacotherapy to Enhance Weight Loss Following Sleeve Gastrectomy
Brief Title: Efficacy of Pharmacotherapy to Enhance Weight Loss Following Sleeve Gastrectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty with enrollment and then Covid pandemic
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HHC-2018-0155
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Metformin; Topiramate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Medication arm (Experimental)
  Interventions: Drug: Administration of weight loss drug (Metformin or Topiramate)
- No medication arm (No Intervention)

INTERVENTIONS:
Drug: Administration of weight loss drug (Metformin or Topiramate) — Patients in this arm will receive either Metformin (500 mg, twice per day) or Topiramate (50 mg, once per day) starting at 4 weeks after laparoscopic sleeve gastrectomy
  Arms: Medication arm

SUMMARY:
The study will investigate the effects of Metformin and Topiramate prescribed at 4 weeks post-surgery on overall weight loss at 6 months post-surgery. The investigators will study patients who, based on current diagnoses and medication regimens, could be expected to benefit the most by taking a medication to facilitate additional post-surgery weight loss. Patients scheduled to undergo laparoscopic sleeve gastrectomy (LSG) at Hartford Hospital's Bariatric and Metabolic Surgery Program will be screened, consented and enrolled in the study. Prior to surgery patients will be randomized to either pharmacotherapy or no pharmacotherapy following LSG. For those randomized to receive pharmacotherapy, medications will be initiated at 4 weeks, as this is the estimated time post-LSG at which patients advance from a liquid diet to soft foods allowing medications to be better tolerated. Once randomly assigned to the medication group, patients will receive Metformin or Topiramate based upon physician judgment and medical history. Dosages will not be adjusted during the course of the study. The primary outcome will be % total body weight loss (%TWL) at 6 months following surgery, as the majority of the weight loss after LSG occurs during the first 6 months. Data collected through up to 12 months will be analyzed. The %TWL for both arms of the study will also be assessed at 8 weeks, 16 weeks, and 9 months and one-year post-LSG. Resolution of comorbidities will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for sleeve gastrectomy as primary bariatric treatment

Exclusion Criteria:

* Qualified for Roux en Y gastric bypass
* On FDA approved weight loss medications prior to bariatric surgery
* Required to continue Topiramate, Zonisamide, and Buproprion for other chronic diseases after bariatric surgery
* On Metformin, Dulaglutide, Exenatide, Exenatide Extended Release, Liraglutide, Empaglifozin, Canaglifozin, Dapaglifozin, Buproprion, Zonisamide, and Topiramate, prior to surgery.
* Have had lap band or other prior bariatric surgery
* Glomular filtration rate < 45
* Over 70 years old
* Not fluent in English

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Weight loss percentage | one year
  Percent of total body weight lost

SECONDARY OUTCOMES:
Rate of Diabetes Resolution | One year
  Resolution of diabetes will be ascertained from the medical chart
Rate of High blood pressure resolution | One year
  Resolution of high blood pressure will be ascertained from the medical chart
Rate of High cholesterol resolution | One year
  Resolution of high cholesterol will be ascertained from the medical chart
Rate of GERD resolution | One year
  Resolution of GERD will be ascertained from the medical chart
Rate of Sleep apnea resolution | One year
  Resolution of sleep apnea will be ascertained from the medical chart

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No